CLINICAL TRIAL: NCT01442532
Title: A Double-Blind, Randomized, Single- and Multiple-Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-38518168 in Japanese and Caucasian Healthy Adult Male Subjects and an Open-Label Drug-Drug Interaction Study to Evaluate the Effect of JNJ-38518168 on the Pharmacokinetics of Midazolam, a CYP3A4 Substrate
Brief Title: A Study of the Safety and Pharmacokinetics of JNJ-38518168 in Japanese and Caucasian Male Participants and the Effect of JNJ-38518168 on the Blood Levels of Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100669; 38518168ARA1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-09-27; First posted 2011-09-28 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Male Volunteer
Keywords: Healthy male volunteer; JNJ-38518168; Midazolam
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: JNJ-38518168 (30 mg)
- 2 (Experimental)
  Interventions: Drug: JNJ-38518168 (10 mg)
- 3 (Experimental)
  Interventions: Drug: JNJ-38518168 (3 mg)
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo
- 5 (Experimental)
  Interventions: Drug: Midazolam and JNJ-38518168

INTERVENTIONS:
Drug: JNJ-38518168 (30 mg) — Type=range, unit=mg, number=30, form=tablet, route=oral use, in single and multiple doses for 14 days
  Arms: 1
Drug: JNJ-38518168 (10 mg) — Type=range, unit=mg, number=10, form=tablet, route=oral use, in single and multiple doses for 14 days
  Arms: 2
Drug: JNJ-38518168 (3 mg) — Type=range, unit=mg, number=3, form=tablet, route=oral use, in single and multiple doses for 14 days
  Arms: 3
Drug: Placebo — Form=tablet, route=oral use, for 14 days
  Arms: 4
Drug: Midazolam and JNJ-38518168 — Midazolam: Type=exact, unit=mg, number=2.5, form=oral solution; route=oral use, on Days 1 and 15; JNJ-38518168: Type=exact, unit=mg, number=30, form=tablet, route=oral use, once daily from Day 2 through Day 15
  Arms: 5

SUMMARY:
The purpose of Part 1 of this study is to evaluate the safety, tolerability, and pharmacokinetics ("PK", how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time) of JNJ-38518168 in comparison with placebo following single dose and 14 days of consecutive dosing in healthy Japanese and Caucasian adult male participants. Part 2 of this study will evaluate the effect of JNJ-38518168 on the pharmacokinetics of midazolam in healthy participants.

DETAILED DESCRIPTION:
Participants will be assigned to either Part 1 or Part 2 of this study. Part 1 will be a single-center, double-blind (participants and study personnel will not know the identity of the treatments), randomized (treatment will be assigned by chance), single- and multiple-dose study. There will be 3 groups in Part 1, and the dosing will be as follows: Group A will receive a single oral dose of 30 mg JNJ-38518168 (given as three 10-mg tablets of JNJ-38518168) or placebo (a treatment identical in appearance to JNJ-38518168 but not containing active drug) (Period 1), and multiple oral doses of 30 mg JNJ 38518168 (given as three 10-mg tablets of JNJ-38518168) or matching placebo once daily for 14 consecutive days (Period 2); Group B will receive a single oral dose of 10 mg JNJ-38518168 or placebo (Period 1), and multiple oral doses of 10 mg JNJ-38518168 or placebo once daily for 14 consecutive days (Period 2); and Group C will receive a single oral dose of 3 mg JNJ-38518168 or placebo (Period 1), and multiple oral doses of 3 mg JNJ-38518168 or placebo once daily for 14 consecutive days (Period 2). At least a 20-day washout period will separate the dose administration in Period 1 and the first dose administration of Period 2. The duration of Part 1 will be approximately 78 days. Part 2 of this study will be a single-center, open-label (participants and study personnel will know the identity of the treatments), non-randomized, multiple dose, drug-drug interaction study. Eligible participants will receive a single oral dose of 2.5 mg of midazolam as oral solution on Day 1, three 10-mg tablets of JNJ-38518168 (30 mg) once daily for 14 consecutive days (Day 2 through Day 15); and another single oral dose of 2.5 mg midazolam on Day 15. The duration of Part 2 of the study will be approximately 42 days. Following an interim safety and PK data analysis, one additional treatment group may be studied to evaluate the effect of JNJ-38518168 at a dose lower than 30 mg once daily on the PK of midazolam. During Parts 1 or 2, participants may be admitted to the clinical unit for periods of up to 7 and 18 days, and follow-up return visits to the clinic will also be required.

ELIGIBILITY:
Inclusion Criteria:

Part 1 only:

* Male, 20 to 55 years of age.
* Be either:
* Of Japanese descent who has resided outside of Japan for no more than 5 years and whose parents and maternal and paternal grandparents are Japanese, as determined by participant's verbal report. Japanese participants must have a valid Japanese passport.

or

* A non-Hispanic Caucasian participant who has Caucasian parents as determined by participant's verbal report.
* Have a body mass index (BMI) of 18.5 kg/m2 to 25 kg/m2 for participants of Japanese descent and between 18.5 kg/m2 and 30 kg/m2 for Caucasian participants.
* Have a body weight of not less than 50 kg.

Part 2 only:

* Male, 18 to 55 years of age
* Have a BMI of 18.5 kg/m2 to 30 kg/m2 and have a body weight of not less than 50 kg.

For both Parts 1 and 2:

* Be otherwise healthy with no clinically significant abnormalities as determined by medical history, physical examination, blood chemistry assessments, hematologic assessments, coagulation and urinalysis, measurement of vital signs, and ECG. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judge the abnormalities or deviations from normal to be not clinically significant.
* If a man is heterosexually active with a woman of childbearing potential, he must be surgically sterile or agree to use a double-barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug.
* Have a blood pressure measurement between 90 and 140 mmHg systolic, inclusive, and between 50 and 90 mmHg diastolic, at screening.
* Have a 12-lead ECG consistent with normal cardiac conduction and function at screening.
* Non-smoker.

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results.
* History of hypersensitivity to or intolerance of midazolam (Part 2 only)
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or admission to the study center in Period 1 as deemed appropriate by the investigator.
* Clinically significant abnormal physical examination, vital signs, or 12-lead ECG at screening or admission to the study center in Period 1 as deemed appropriate by the investigator.
* Has any known malignancy or a history of malignancy (with the exception of basal cell carcinoma, squamous cell carcinoma in situ of the skin, or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years prior to the first administration of study drug).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The number of Japanese participants with adverse events | Up to 10 weeks
Blood tests in Japanese participants | Up to 10 weeks
Clinical laboratory tests in Japanese participants | Up to 10 weeks
Electrocardiograms in Japanese participants | Up to 10 weeks
Blood levels of JNJ-38518168 in all participants | Up to 10 weeks

SECONDARY OUTCOMES:
The number of Caucasian participants with adverse events | Up to 10 weeks
Blood tests in Caucasian participants | Up to 10 weeks
Clinical laboratory tests in Caucasian participants | Up to 10 weeks
Electrocardiograms in Caucasian participants | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC & Development, L.L.C., Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Cypress, California, United States